CLINICAL TRIAL: NCT00639041
Title: Changes in Blood Lipids After Long Time Consumption of n-3 LC-PUFA-enriched Dairy Products in Hypertriglyceridemic Patients: a Randomized, Double-blind, Cross-over Study
Brief Title: Changes in Blood Lipids After Long-term Consumption of n-3 LC-PUFA-Enriched Dairy Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: LSEP H26_06; Gerhard.Jahreis@uni-jena.de
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2008-02

CONDITIONS: Hypertriglyceridemia
Keywords: n-3 LC-PUFA; hypertriglyceridemic; human; TAG
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- n-3 LC-PUFA (Active Comparator)
  Interventions: Dietary Supplement: n-3 LC-PUFA

INTERVENTIONS:
Dietary Supplement: n-3 LC-PUFA — n-3 LC-PUFA supplemented dairy products (yoghurt, cheese, butter): 3.3 g n-3 FA/d
  Arms: n-3 LC-PUFA
Dietary Supplement: Placebo — dairy products without special oils
  Arms: placebo

SUMMARY:
The study was performed to investigate the effects of n-3 LC-PUFA supplemented dairy products cardiovascular risk factors in hypertriglyceridemic patients.

DETAILED DESCRIPTION:
Recent studies suggest that n-3 LC-PUFA intake might be useful to prevent coronary heart diseases.

As a precondition for participating in this study, the patients were provided information in writing and verbally about the details of the study. Informed consent was obtained from all volunteers. Before the beginning of the study, all participants were subject to a medical examination by their general practitioners. Fifty-one hypertriglyceridemic patients (25 f, 26 m; with triacylglyceride (TAG) values ≥ 150 mg/dl or ≥ 1.7 mmol/L) entered the study.

The placebo-controlled, randomized double-blind cross-over study consisted of two investigation periods of 15 weeks, with a ten-week washout period in between. After the washout period the intervention was crossed between the groups and the respective products were consumed for another 15 weeks. Patients received about 40 g fat daily (200 g yoghurt with 3.8% fat, 30 g cheese with about 50% fat in the dry matter, and 20-30 g butter). The milk fat was partially exchanged by special oils (fish oil, rapeseed oil) with high amounts of eicosapentaenoic acid (EPA), docosahexaenoic acid (DHA), and alpha linolenic acid (ALA). The daily dose of n-3 FA amounted to 3.3 g, consisting of 1.5 g EPA, 1.2 g DHA, 0.2 g DPA, and 0.2 g ALA.

Venous blood and 24h urine were collected at the beginning and at the end of each period.

ELIGIBILITY:
Inclusion Criteria:

* TAG values ≥ 150 mg/dl or ≥ 1.7 mmol/L

Exclusion Criteria:

* blood diluted medications
* lipid lowering medications
* glucocorticoids
* gastrointestinal or metabolic diseases (e.g., diabetes mellitus, hyperthyroidism or hypothyroidism, hypercholesteremic patients with familial previous impacts)
* daily alcohol abuse
* taking dietary supplements (e. g., fish oil capsules, vitamin E)
* known allergies or foodstuff indigestibility

Ages: 43 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
blood lipids (total cholesterol, high density cholesterol (HDL), low density cholesterol (LDL), TAG) | 15 weeks

SECONDARY OUTCOMES:
blood pressure | 15 weeks
fibrinogen | 15 weeks
homocysteine | 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Jahreis, Prof. Dr., Principal Investigator — University of Jena, Dept. of Nutritional Physiology
Locations (1):
- Facility: University of Jena, Institute of Nutrition, Department of Nutritional Physiology, Jena, Thuringia, Germany

REFERENCES:
- [Background] Dawczynski C, Martin L, Wagner A, Jahreis G. n-3 LC-PUFA-enriched dairy products are able to reduce cardiovascular risk factors: a double-blind, cross-over study. Clin Nutr. 2010 Oct;29(5):592-9. doi: 10.1016/j.clnu.2010.02.008. Epub 2010 Mar 20. PMID 20304540